CLINICAL TRIAL: NCT06041737
Title: Determination of a Profile of Patients with Renal Failure to Be Supported As a Priority in the Care Pathway in Order to Avoid Emergency Hospitalizations.
Acronym: DETERPROFIPA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/0023
Record Dates: First submitted 2023-09-11; First posted 2023-09-18 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Renal Failure
Keywords: Chronic kidney disease; Patients profile; Hospitalization profile; Advanced practice nurse; Organizational protocol
MeSH Terms: conditions — Renal Insufficiency; Renal Insufficiency, Chronic | interventions — Referral and Consultation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: consultation — nephrology consultation during 2020

SUMMARY:
The purpose of this study is to map the population of stage 4 and 5 kidney failure patients followed in consultation by the CHSF nephrology team and to determine the factors associated with recurrent hospitalizations.

DETAILED DESCRIPTION:
This observational study on retrospective data does not justify a specific calculation of numbers. Over the 27-month observation period, have been identified in the department an active file of approximately 440 stage 4 or 5 chronic kidney failure patients eligible for the study.

The qualitative variables will be expressed in numbers and corresponding percentages, and compared by Fisher's exact test. Quantitative variables will be expressed by their mean and standard deviation or by their median and interquartiles, depending on their distribution. They will be compared by the Student test in the case of a normal distribution, by the Wilcoxon test otherwise.

The main outcome criterion, namely the occurrence of hospitalization during the observation period, will be analyzed using a logistic regression model. The covariates tested in the model will be :

* Age
* Gender
* Helpers among: Parent, Sibling, Child, Spouse, neighbors, friend, Social care (social security (SSC), mutual insurance or universal health coverage (CMU)
* Active, disabled, retired
* MRC Stage (4 or 5) in 2020
* Mode of entry into nephrology consultation (after hospitalization in Nephrology, attending physician, diabetologist, cardiologist, other)
* History and associated comorbidities including high blood pressure, diabetes, dyslipidemia, vascular pathologies, heart disease, sleep apnea syndrome, obesity, other chronic pathologies.
* Number of chronic pathologies of the patient
* The pathology(s) retained by the nephrologist as responsible for the kidney disease (several pathologies can be retained and reported as such)
* Number of treatments on the patient's prescription
* Treatments: hypotensive, antidiabetic, hypolipidemic, diuretic, potassium chelator, cardiac treatment, antithrombotics, others
* Number of years of follow-up in nephrology at the CHSF before the period studied.
* Status of known patients at the end of follow-up (it can be before 03/31/2022 if the patient has moved to another status before) among: consultation, dialysis (urgent or normal), transplant, death, lost to follow-up .
* Did the patient benefit from pre-dialysis information, at what Glomerular Filtration Rate (GFR) and what was his choice (peritoneal dialysis, hemodialysis or conservative treatment)
* Did the patient benefit from an arteriovenous fistula, at what GFR
* Did the patient benefit from a pre-transplant assessment
* The number of consultations by a nephrologist, in consultation or in day hospital.
* The number of consultations canceled by the patient.
* The number of consultations not honored by the patient.
* Le nombre de consultations sans bilan récent.
* The GFR at the consultation
* Unscheduled hospitalizations at the CHSF during follow-up, whether in nephrology or in another hospital department.
* The reason(s) for unscheduled hospitalizations related to renal pathology (cardiac decompensation, anemia, sodium and water overdose, acute lung edema (APO), high blood pressure (hypertension), emergency dialysis starts, renal failure acute (ARI), and ionic disorders,)
* The number of days for each hospitalization. The log-linearity of the quantitative variables will be evaluated by graphical method. In the event of non-log-linearity, the variable will be discretized according to its median or according to the inflection points of the curve. Covariates whose unadjusted Odds Ratio has a p value less than 0.20 will be retained in the multivariate model. All second-order interactions will be tested. Multicollinearity phenomena will be evaluated by measuring variance inflation factors, with a positivity threshold set at 2.5. A variable selection using a descending step-by-step method minimizing the Akaiké criterion will then be carried out. The area under the ROC curve of the final model as well as the p value of the Hosmer-Lemeshow test will be specified.

In secondary analyses, patients who were not hospitalized during the observation period will be compared to those who had 1 to 3 hospitalizations and to those who had 4 or more hospitalizations. Qualitative variables will be analyzed using Fisher's exact test. The quantitative variables will be compared by analysis of variance if its conditions of application are met, by the Kruskal-Wallis test otherwise. In the event of significance, comparisons 2 by 2 will be carried out, respectively by the Student test or the Wilcoxon test, with adjustment of the value of p by the Bonferroni-Holm correction in order to take account of the multiple comparisons.

All the tests will be carried out bilaterally, with a 1st type risk set at 5%. The analysis will be performed using R software (version 4.3.1 © 2023 The R Foundation for Statistical Computing).

Management of missing data:

no plan to replace missing data for this observational data study, the design of which in any case makes the presence of missing data in numbers unlikely, particularly concerning the main criterion.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* patients with stage 4 or 5 kidney failure who had at least one nephrology consultation during 2020.

Exclusion Criteria:

- Patients informed of the study who objected to the collection of their data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with renal insufficiency in stage 4 or 5 having had at least one nephrology consultation at the CHSF during the year 2020.
Sampling Method: Non-Probability Sample
Enrollment: 405 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Determination of factors associated with recurrent hospitalizations in patients followed for stage 4 or 5 Chronic Renal Failure. | at day 0
  characteristics of patients who have had at least one hospitalization and those who have never been hospitalized over the period from January 1, 2020 to March 31, 2022

SECONDARY OUTCOMES:
Mapping of the population of patients with stage IV and V renal failure followed in consultation by the CHSF nephrology team. | at day 0
  General and medical characteristics of patients followed at the CHSF in nephrology consultation for stage 4 or 5 CKD
Determination of the profile(s) of stage 4 or 5 CKD patients with recurrent hospitalizations. | at day 0
  Comparison of patient cohorts with a single hospitalization and more than 4 hospitalizations

CONTACTS AND LOCATIONS:
Overall Officials: Christine BOUHELIER, nurse, Principal Investigator — Centre Hospitalier Sud Francilien
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France

IPD SHARING:
Plan to Share IPD: No